CLINICAL TRIAL: NCT02724930
Title: Cooperative Pain Education and Self-management
Acronym: COPES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Connecticut Healthcare System (U.S. Federal Agency)
Collaborators: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 0012
Record Dates: First submitted 2016-03-22; First posted 2016-03-31 (Estimated); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Chronic Low Back Pain
Keywords: low back pain, chronic pain, cognitive behavior therapy
MeSH Terms: conditions — Low Back Pain; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Implementation (No Intervention): Standard COPES implementation consists of provider education including brief in-person presentations and written material.
- Implementation Facilitation (Experimental): Enhanced facilitation of COPES implementation.
  All clusters start in the standard implementation group and cross-over from the control group to the intervention group in a randomized stepped-wedge fashion at 7 time points over the course of the 33 week implementation.
  Interventions: Behavioral: Enhanced facilitation of COPES

INTERVENTIONS:
Behavioral: Enhanced facilitation of COPES — Enhanced facilitation of COPES implementation consists of promotional meetings, automated case finding and proactive outreach to recruit patients, marketing and educational materials, local champion, and academic detailing.
  Arms: Implementation Facilitation

SUMMARY:
This study will test the effectiveness of using enhanced facilitation strategies on implementation of an automated Interactive Voice Response (IVR) system as a means to remotely deliver in-home self-management support to Veterans with chronic pain. The implementation intervention uses an enhanced facilitation approach paired with automated case finding and direct patient outreach to encourage uptake of Cooperative Pain Education and Self-management (COPES). A nested effectiveness study will measure pre-post differences in pain-relevant outcomes (pain intensity, physical functioning and physical activity). The investigators will use a stepped wedge cluster design in which clusters will be randomized to the timing of the introduction of enhanced COPES implementation. Investigators will assess the efficacy of the facilitation based implementation strategy by evaluating COPES uptake in the implementation settings.

DETAILED DESCRIPTION:
Cognitive behavioral therapy (CBT) for chronic pain is a commonly used evidence-based self-management intervention. Though effective, CBT requires that patients attend multiple in-person visits and that highly trained staff be available to provide care. For these reasons CBT is resource intensive, often inaccessible to Veterans, and delivered unevenly across patients and facilities. In a Veterans Health Administration Office of Health Services Research and Development (HSR&D) IIR-funded trial, investigators found that CBT delivered primarily via an automated Interactive Voice Response (IVR) system (Cooperative Pain Education and Self-management or COPES) leads to patient-centered outcomes that are comparable to standard United States Department of Veterans Affairs (VA) approaches in which CBT is delivered in-person by a therapist over ten weekly sessions. In this study, implementation facilitation will be guided by the Consolidated Framework for Implementation Research (CFIR) which provides a set of constructs to identify potential barriers and facilitators to implementation. The primary objective of this project is to evaluate the effectiveness of the facilitation approach paired with automated case finding and direct patient outreach on uptake of COPES in the clinical care setting. Study investigators will specifically target Veterans who receive care at community-based outpatient clinics (CBOCs) because these sites typically have few or no therapists trained in CBT for chronic pain.

Description of COPES: COPES is a 10-week, IVR-facilitated program of CBT for chronic pain. The primary components of COPES include: 1) a self-help handbook to teach Veterans pain self-management skills and describe the weekly skill practice goals, 2) a pedometer-facilitated progressive walking program (all COPES patients will be given an Omron Go Smart, Model HJ-112 pocket pedometer at the time of enrollment), and 3) daily, automated IVR calls to collect patient-reported pain intensity and pain-related interference, sleep quality, pedometer-measured step count, and adherence to the pain coping skill practice ratings. Participants will also receive a weekly, two to four minute pre-recorded, personalized therapist message via the IVR system based on the participant's IVR-recorded data. Therapists provide feedback on the participant's weekly average pain intensity, sleep, steps, and pain coping skill practice, note any changes from the prior week, and comment on symptom or activity patterns. Therapists also provide reinforcement for goal accomplishment, help patients make connections among pain, pain coping skill practice, and goal accomplishment, and assign a steps and skill practice goal for the upcoming week.

Research Design: Study investigators will test the effectiveness of the facilitation approach to implement COPES as a means to remotely deliver in-home self-management support to Veterans with chronic pain. To evaluate the implementation's success, study investigators will conduct a multi-site, stepped wedge, Hybrid III trial in 17 CBOCs affiliated with three geographically dispersed sites (VA Boston, VA Palo Alto, and Roudebush VA in Indianapolis). Clusters (k=17 CBOCs) will be randomized to 6 different time periods proportional to approximate eligible patient population size. Each CBOC will serve as its own control for a period of time before "transitioning" into enhanced facilitation; the time of this transition is randomized in a stepped fashion. The primary outcome for evaluating implementation success will be patient enrollment in COPES. The secondary outcome will be provider referral. Other outcomes that will be investigated as part of the nested COPES effectiveness study will be Veterans' physical functioning, pain intensity, and physical activity.

Methodology: Study investigators will evaluate the success of the implementation strategy by evaluating the proportion of patients who are offered enrollment in COPES who actually enroll. Additionally, study investigators will conduct a formative evaluation to inform, refine and evaluate implementation of COPES. The evaluation will include interviews with VA staff and patients with chronic back pain at the proposed implementation sites. Interview guides will be based on CFIR model constructs using questions adapted from the CFIR interview guide. Investigators will also measure pre-post differences in pain-relevant outcomes (pain intensity, physical functioning and physical activity).

ELIGIBILITY:
Inclusion Criteria:

Veterans COPES:

1. Back-pain-related International Classification of Diseases (ICD)-9 diagnosis
2. Pain intensity rating of ≥4 (indicating moderate pain) on the 0-10 Numerical Rating Scale on at least two separate outpatient encounters at a CBOC in the prior year
3. CBOC patient at VA Boston, VA Palo Alto or Roudebush VA

Veterans Interviews:

1. Those who are eligible for COPES, but who have not been asked to enroll (pre-implementation period)
2. Those who participate in COPES (post-implementation)
3. Those who decline enrollment in COPES (post-implementation)
4. CBOC patients at VA Boston, VA Palo Alto or Roudebush VA

Admin, Champion, Provider Interviews:

1. Employed at the project implementation sites

Exclusion Criteria:

Veterans (COPES & Interviews):

1. Diagnosis of cancer, dementia, schizophrenia, and active alcohol or substance abuse
2. Psychiatric hospitalization in the past 30 days
3. Patients who are designated as fall risks and/or have active diabetic foot ulcers

Admin, Champion, Provider Interviews:

1. Not employed at the project implementation sites

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2020-08-27 (Actual); Study Completion 2020-08-27 (Actual)

PRIMARY OUTCOMES:
Patient enrollment | Baseline, 6 months post-facilitation, and study end (up to 30 months)
  Patient enrollment measured as the probability an eligible patient enrolls in Cooperative Pain Education and Self-management (COPES).

SECONDARY OUTCOMES:
Provider referrals | Baseline, 6 months post-facilitation, and study end (up to 30 months)
  Provider referrals to COPES measured as the total number of provider referrals and the number of referrals per provider by: site, time point, and overall.

OTHER OUTCOMES:
Pain-related interference | Baseline, 6 months post-facilitation, and study end (up to 30 months)
  Pain-related interference will be assessed using the interference items of the "PEG 3 A Three-Item Scale Assessing Pain Intensity and Interference" (PEG-3) which assesses interference with general activity and enjoyment of life.
Pain intensity | Baseline, 6 months post-facilitation, and study end (up to 30 months)
  Pain intensity will be assessed using the pain intensity question of the PEG-3.
Physical activity | Baseline, 6 months post-facilitation, and study end (up to 30 months)
  Physical activity will be assessed by pedometer-measured step count.

CONTACTS AND LOCATIONS:
Overall Officials: Alicia A Heapy, PhD, Principal Investigator — VA Connecticut Healthcare System; John D Piette, PhD, Principal Investigator — VA Ann Arbor Healthcare System
Locations (3):
- United States (3):
  - VA Palo Alto Healthcare System, Menlo Park, California
  - Richard L. Roudebush VA Medical Center, Indianapolis, Indiana
  - VA Boston Healthcare System, Brockton, Massachusetts

IPD SHARING:
Plan to Share IPD: No